CLINICAL TRIAL: NCT00559338
Title: Acutely Decompensated Heart Failure in a County Emergency Department: A Double Blind Randomized Controlled Comparison of Nesiritide vs. Placebo Treatment
Brief Title: Impact of Nesiritide Infusion for Decompensated Heart Failure in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB0603-412
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Heart Failure, Congestive; Cardiomyopathy
Keywords: CHF; Heart Failure; Dyspnea; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Dyspnea | interventions — Natriuretic Peptides; Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The intravenous infusion of nesiritide consisted of a bolus dose of 2mcg/kg followed by the infusion rate of 0.01 mcg/kg/min for up to eight hours. The nesiritide was mixed in 250 ml of 0.9% normal saline solution.
  Interventions: Drug: recombinant B-type, natriuretic peptide
- 2 (Placebo Comparator): The intravenous infusion of placebo consisted of a bolus dose of 2mcg/kg followed by the infusion rate of 0.01 mcg/kg/min for up to eight hours. The placebo was mixed in 250 ml of 0.9% normal saline solution.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: recombinant B-type, natriuretic peptide — The intravenous infusion of nesiritide consisted of a bolus dose of 2mcg/kg followed by the infusion rate of 0.01 mcg/kg/min for up to eight hours. The nesiritide was mixed in 250 ml of 0.9% normal saline solution.
  Other Names: Nesiritide
  Arms: 1
Drug: placebo — The intravenous infusion of placebo consisted of a bolus dose of 2mcg/kg followed by the infusion rate of 0.01 mcg/kg/min for up to eight hours. The placebo was mixed in 250 ml of 0.9% normal saline solution.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if an 8hr infusion of nesiritide in the emergency department in the Acutely decompensated heart failure patients will decrease 30 day recidivism.

DETAILED DESCRIPTION:
In view of the high return admission rate to our county ED for heart failure, we hypothesized that our higher risk patient population might realize a decrease in the return admission rate as a benefit from early ED administration of nesiritide. We also acknowledged that the safety of nesiritide in our patient population had not been well established. Thus, we opted to test the hypothesis that an 8-hour ED infusion of nesiritide [in addition to protocol specified standard therapy] in ADHF patients from an urban patient population consisting of predominately African Americans and Hispanics will decrease 30-day readmission rates without provoking harm.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were adults greater than 18 years of age
* A history of established heart failure
* Dyspnea at rest or with minimal exertion and with a respiratory rate greater than 24 breaths per minute
* Evidence of volume overload based on physical exam findings or chest radiograph, and a brain natriuretic peptide (BNP) level greater than 100 pg/ml.

Exclusion Criteria:

* Systolic blood pressure of less than 90 mm Hg
* Frank or impending cardiogenic shock
* Cardiopulmonary arrest
* Evidence of low cardiac output (cold clammy extremities
* Mental status changes)
* New onset congestive heart failure
* Suspected acute coronary syndrome (elevated troponin, New electrocardiographic changes, or history consistent with cardiac ischemia)
* High clinical suspicion of pulmonary embolism
* End-stage renal disease (on dialysis or imminent)
* Active use of nitroglycerin or inotropic infusions in the ED
* Ventricular tachycardia
* Allergy to nesiritide or its components
* Patient not needing intravenously diuretic therapy in the ED
* Normal BNP level
* Inability to follow-up
* Pregnancy or suspected pregnancy; or
* Actively receiving other investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2003-12; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of 30 day readmission to the ED or readmission after an 8-hr infusion of nesiritide, in addition to standard care, compared to placebo plus standard care | 30-day

SECONDARY OUTCOMES:
Secondary outcome measures included admission to the hospital after an 8-hr infusion of nesiritide, return to the ED or readmission at 7 days, 60 days, and 90 days | 90-days

CONTACTS AND LOCATIONS:
Overall Officials: Adam H Miller, Principal Investigator — UT Southwestern Medical Center Dallas
Locations (1):
- Parkland Hospital, Dallas, Texas, United States